CLINICAL TRIAL: NCT06882096
Title: Tracing the Metabolic Flux of Orally Administered NAD+ Precursors in Healthy Young and Older Adults
Brief Title: Tracing the Metabolic Flux of Orally Administered NAD+ Precursors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Metro International Biotech, LLC (Industry)
Responsible Party: Principal Investigator, Shalender Bhasin, Principal Investigator, Metro International Biotech, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MBT-1918/1932-MET
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Nicotinamide Mononucleotide; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMN- Nicotinamide Mononucleotide (Active Comparator): This arm will include 16 participants (8 young and 8 older adults) who will receive NMN once daily for 14 consecutive days.
  Interventions: Drug: Nicotinamide Mononucleotide (NMN)
- NAM- Nicotinamide (Active Comparator): This arm will include 16 participants (8 young and 8 older adults) who will receive NAM once daily for 14 consecutive days.
  Interventions: Drug: Nicotinamide (NAM)

INTERVENTIONS:
Drug: Nicotinamide Mononucleotide (NMN) — Nicotinamide Mononucleotide (NMN)
  Arms: NMN- Nicotinamide Mononucleotide
Drug: Nicotinamide (NAM) — Nicotinamide (NAM)
  Arms: NAM- Nicotinamide

SUMMARY:
We are doing this research to learn how healthy younger and older adults use two forms of vitamin B3-called nicotinamide mononucleotide (NMN) and nicotinamide (NAM)-to make NAD+. NAD+ is a natural substance that cells need for energy and other important processes. Our goal is to find out how these NAD precursors are absorbed and metabolized and how they raise NAD+ in different tissues.

Who can join? Healthy adults men and women aged 18 to 40 (younger group) or 65 and older (older group) Participants with a body mass index ranging between 19 and 35 No major health issues like diabetes or severe kidney disease

What will happen? Participants will take labeled or unlabeled NMN or NAM by mouth every day for 14 days.

Researchers will collect blood, urine, and stool samples. Researchers also do a small muscle biopsy (under local numbing) twice to check how these NAD precursors raise NAD+ in muscle.

Why is this important? NAD+ levels may drop as people age, and this drop could affect overall health and energy in cells.

A better understanding of how NMN and NAM are metabolized in the body to raise NAD+ levels in both younger and older adults may help us optimize dosing and strategies for raising NAD in older people.

Possible benefits and risks:

Participants may not get any direct health benefit from this study; the main goal is to gather new knowledge.

NMN and NAM appear safe in the doses used. A muscle biopsy may cause soreness or bruising.

Researchers will monitor participants closely for any side effects throughout the study.

DETAILED DESCRIPTION:
Background and Significance

1.1 Role of NAD+ in Physiology Nicotinamide adenine dinucleotide (NAD+) is a key coenzyme in all living organisms, existing in oxidized (NAD+) and reduced (NADH) forms. Beyond its vital role in redox reactions and ATP generation, NAD+ also serves as a co-substrate for several signaling enzymes such as sirtuins, PARPs, and CD38. Systemic NAD+ insufficiency can cause diseases like pellagra; reduced NAD+ availability has been implicated in aging and age-related disorders.

1.2 Oral NAD+ Precursors Administration of NAD+ precursors (e.g., NMN, NR, NAM) can boost NAD+ levels. Although human research has shown that oral NMN raises blood NAD+ concentrations, many aspects of its absorption, metabolism, and overall bioavailability are still poorly understood. Rodent studies suggest oral NMN undergoes extensive first-pass metabolism in the gut, with partial conversion to NAM prior to entering systemic circulation.

1.3 Aging and NAD+ In rodent models, NAD+ levels frequently decline as the animals get older. Some evidence indicates that NAD+ turnover may be elevated in aging rodents, suggesting a higher rate of NAD+ consumption. However, equivalent tracer studies have not yet been conducted in humans.

1.4 Need for Human Tracer Studies These compounds are being investigated for the prevention and treatment of age-related diseases. There is a need to clarify how they are absorbed and how exactly they elevate NAD+ in different tissues. Using stable isotope-labeled NMN and NAM will help map the flux from oral precursors into blood, muscle, urine, and stool, and will also reveal how aging influences NAD+ turnover.

2. Aims and Objectives

Aim 1: Use stable isotope tracers and mass spectrometry in healthy young adults to track how orally administered NMN or NAM are metabolized, how they enter NAD+ pools, and how much is excreted or converted to other metabolites.

Aim 2: Compare these same fluxes in older adults (≥65 years). Investigators specifically want to see whether age alters the metabolic route from precursor to NAD+ and whether older adults exhibit higher consumption (turnover) of NAD+.

3. Study Design

3.1 Overview Single-center trial at Brigham and Women's Hospital.

Groups: Two main groups of participants:

Group A (NMN group): 16 participants (8 young adults aged 18-40; 8 older adults aged ≥65).

Group B (NAM group): 16 participants (8 young; 8 older). Each participant takes either NMN or NAM orally for 14 days. The study uses stable isotopes (non-radioactive) to label NMN or NAM in order to track how these molecules appear in NAD+ and its downstream metabolites.

3.2 Treatment Duration Participants receive daily doses of their assigned treatment (NMN or NAM) for 14 days. Detailed sampling done on Days 1 and 14.

3.3 Dosage NMN: 1000 mg once daily (four 250 mg capsules). NAM: 370 mg once daily. On Days 1 and 14, the entire oral dose is fully labeled with stable isotopes; on the intermediate days (2-13), the product is unlabeled.

3.4 Key Assessments Blood draws at multiple time points (e.g., pre-dose, 30 min, 1 hr, 2 hr, 4 hr, 8 hr) on Days 1 and 14.

Muscle biopsies of the vastus lateralis (Days 1 and 14, typically ~6-8 hours after dose) to determine how much labeled precursor appears in muscle NAD+ pools.

Timed Collection of urine and stool on Days 1-2 and 14-15 to see how the precursor or NAD+ metabolites are excreted and to characterize gut microbiome (which can influence NAD+ precursor metabolism and may be affected by NMN or NAM).

4. Endpoints

Primary Endpoints (for NMN group) Fraction of peripheral blood NAD+ containing the stable isotope labelled tracer

Primary Endpoints (for NAM group) Fraction of peripheral blood NAD+ containing the stable isotope labelled tracer

5. Study Procedures Screening Phase (up to 4 weeks before Day 1) Medical history, demographics, laboratory tests (CBC, chemistry, A1C), physical exam, and EKG if indicated.

Confirm eligibility. Intervention Phase (Days 1-14)

Day 1:

Collect baseline blood samples and muscle biopsy. Blood draws at multiple time points (e.g., pre-dose, 30 min, 1 hr, 2 hr, 4 hr, 8 hr).

Administer stable-isotope-labeled product (NMN or NAM) at time 0. Repeat blood draws at specified intervals. Collect urine and stool.

Day 2:

Additional blood draws. Begin taking unlabeled study product daily at home.

Days 3, 5, 8:

Short visits for blood sampling, vital signs, adherence check.

Day 14:

Collect baseline blood samples and muscle biopsy. Blood draws at multiple time points (e.g., pre-dose, 30 min, 1 hr, 2 hr, 4 hr, 8 hr).

Administer stable-isotope-labeled product (NMN or NAM) at time 0. Collect urine and stool.

Day 15:

Unlabeled Treatment (NAM or NMN) administration. Follow-up blood draws.

Follow-up Phase:

Days 16, 43:

Final safety labs, check for adverse events, measure any labeled/unlabeled NAD+ or metabolites that might linger.

6. Risks and Safety

Drug Safety:

Previous Phase 1 trials show 1000 mg NMN up to twice daily is safe and well-tolerated, with no serious drug-related adverse events.

NAM is generally recognized as safe at these doses. High-dose niacin can cause flushing, GI disturbance, or liver enzyme elevations, but those have not been seen with NMN or NAM.

Muscle Biopsy:

Potential for temporary discomfort, bruising, or rare infection at the biopsy site. The team will use local anesthetic and standard sterile technique.

Blood Draws:

Common risks include transient pain or bruising, and rarely infection.

Urine and Stool Collection:

Main risk is inconvenience and mild discomfort; no significant medical risk from the collection itself.

Adverse Events Reporting:

The protocol specifies regular monitoring and reporting. A Safety Review Committee (SRC) meets every six months.

7. Statistical Analysis

Primary Analyses:

Quantify the fraction of labeled NAD+ vs. unlabeled in blood, PBMCs, muscle, urine, and stool.

Compare young vs. older adults to see whether aging shifts the route or magnitude of NAD+ precursor metabolism.

Models:

Mixed-model repeated measures (MMRM) or ANCOVA with factors for age, sex, and baseline values.

Sample Size:

16 subjects per arm (8 young + 8 older in NMN group; 8 young + 8 older in NAM group) is based on pilot data and the specialized nature of stable-isotope tracing.

8. Study Conduct and Logistics

Randomization:

1:1 ratio to NMN vs. NAM, block-randomized, stratified by age group.

Blinding:

The protocol is an open-label comparison of two labeled precursors.

Data Management:

Electronic CRFs, redcap database, verification by investigators.

Monitoring:

Internal team plus sponsor oversight.

Ethical Considerations:

IRB approval, informed consent detailing objectives, procedures, and risks. Emphasis on ensuring participant safety.

9. Importance and Potential Impact

The protocol addresses critical gaps in knowledge like how orally ingested NAD+ precursors (NMN, NAM) become NAD+ in human tissues.

Results will inform whether older adults have distinctly higher NAD+ turnover and might respond differently to NAD+ augmentation.

Findings could shape clinical dosing recommendations for NMN/NAM in therapeutic or preventive settings related to aging and metabolic health.

ELIGIBILITY:
INCLUSION CRITERIA

A participant may be enrolled if he/she is:

1. A healthy, community-living, man or a woman between 18 and 40 years, inclusive or 65 years or older
2. Has a body mass index (BMI) between 19 and 35 kg/m2, inclusive
3. Is free from clinically significant medical problems as determined by the Investigator
4. Is capable of providing written informed consent.
5. Is willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act.

EXCLUSION CRITERIA

A subject may not be enrolled if s/he:

1. Has AST or ALT > 2 times the upper limit of normal
2. Hematocrit < 36% or > 51% for men, or < 35% to > 48% for women
3. Diagnosis of diabetes, using diabetes medications or an A1C > 6.4%
4. Serum creatinine > 2.0 mg/dL or eGFR <60 mL/min
5. Prohibited medications and substances: use of anabolic steroids, rhGH, DHEA, androstenedione, or any performance enhancing drug; Current use of opiates, amphetamine, cannabinoids and cocaine
6. Use of any dietary supplement. Subjects who are using a supplement containing NAM (or niacin or NMN or NR) may be included if they agree to stop supplement at least 2 weeks before randomization.
7. For women only: Pregnant or planning to get pregnant over the next 6 months, or lactating
8. Participation in an investigational trial within the past 3 months
9. Other medical conditions which, in the opinion of the investigator, would jeopardize safety or impact the validity of the study results

For women only:

Female of childbearing age: Use of oral contraceptives is allowed provided the contraceptive regimen was initiated at least 3 months before randomization and the participant agrees not to change the regimen during the course of the study.

Excluded Medications and Treatments

1. The ingestion of the following is prohibited during 14 days prior to Day 0 and for the duration of the intervention period:

   * Products that contain niacin, nicotinic acid, nicotinamide in any form, other than natural foods
   * Herbal supplements
2. Treatment with another investigational drug, investigational device, or approved therapy for investigational use within 3 month is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Labelled NAD+ in Peripheral Blood | During the Study Intervention Period Day 1 through Day 14
  Quantify the fraction of peripheral blood. NAD+ containing the stable isotope labelled tracer

SECONDARY OUTCOMES:
Labelled NAD+ in Muscle | During the Study Intervention Period Day 1 through Day 14
  Quantify the fraction of muscle NAD+ containing the stable isotope labelled tracer
1-Methyl nicotinamide (MeNAM) in Plasma | During the Study Intervention Period Day 1 through Day 14
  Measure the labelled reading of Plasma NAD+ metabolite 1-Methyl nicotinamide (MeNAM)
1-Methyl nicotinamide (MeNAM) in Muscle | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Muscle NAD+ metabolite 1-Methyl nicotinamide (MeNAM)
1-Methyl nicotinamide (MeNAM) in Urine | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Urine NAD+ metabolite 1-Methyl nicotinamide (MeNAM)
1-Methyl nicotinamide (MeNAM) in Stool | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Stool NAD+ metabolite 1-Methyl nicotinamide (MeNAM)
N-methyl-2-pyridone-5-carboxamide (2PY) in Plasma | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Plasma metabolite N-methyl-2-pyridone-5-carboxamide (2PY)
N-methyl-2-pyridone-5-carboxamide (2PY) in Muscle | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Muscle NAD+ metabolite N-methyl-2-pyridone-5-carboxamide (2PY)
N-methyl-2-pyridone-5-carboxamide (2PY) in Urine | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Urine NAD+ metabolite N-methyl-2-pyridone-5-carboxamide (2PY)
N-methyl-2-pyridone-5-carboxamide (2PY) in Stool | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Stool NAD+ metabolite N-methyl-2-pyridone-5-carboxamide (2PY)
Nicotinamide in Plasma | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Plasma NAD+ metabolite- Nicotinamide
Nicotinamide in Muscle | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Muscle NAD+ metabolite Nicotinamide
Nicotinamide in Urine | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Urine NAD+ metabolite Nicotinamide
Nicotinamide in Stool | During the Study Intervention Period Day 1 through Day 14
  Measure the labeled reading of Stool NAD+ metabolite Nicotinamide

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MB, BS, Principal Investigator — Brigham and Women's Hosptial
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauve AA, Wang Q, Zhang N, Kang S, Rathmann A, Yang Y. Triple-Isotope Tracing for Pathway Discernment of NMN-Induced NAD+ Biosynthesis in Whole Mice. Int J Mol Sci. 2023 Jul 5;24(13):11114. doi: 10.3390/ijms241311114. PMID 37446292
- [Background] Amjad S, Nisar S, Bhat AA, Shah AR, Frenneaux MP, Fakhro K, Haris M, Reddy R, Patay Z, Baur J, Bagga P. Role of NAD+ in regulating cellular and metabolic signaling pathways. Mol Metab. 2021 Jul;49:101195. doi: 10.1016/j.molmet.2021.101195. Epub 2021 Feb 17. PMID 33609766
- [Background] Pencina KM, Lavu S, Dos Santos M, Beleva YM, Cheng M, Livingston D, Bhasin S. MIB-626, an Oral Formulation of a Microcrystalline Unique Polymorph of beta-Nicotinamide Mononucleotide, Increases Circulating Nicotinamide Adenine Dinucleotide and its Metabolome in Middle-Aged and Older Adults. J Gerontol A Biol Sci Med Sci. 2023 Jan 26;78(1):90-96. doi: 10.1093/gerona/glac049. PMID 35182418
- [Background] Pencina KM, Valderrabano R, Wipper B, Orkaby AR, Reid KF, Storer T, Lin AP, Merugumala S, Wilson L, Latham N, Ghattas-Puylara C, Ozimek NE, Cheng M, Bhargava A, Memish-Beleva Y, Lawney B, Lavu S, Swain PM, Apte RS, Sinclair DA, Livingston D, Bhasin S. Nicotinamide Adenine Dinucleotide Augmentation in Overweight or Obese Middle-Aged and Older Adults: A Physiologic Study. J Clin Endocrinol Metab. 2023 Jul 14;108(8):1968-1980. doi: 10.1210/clinem/dgad027. PMID 36740954
- [Background] Dutta T, Kapoor N, Mathew M, Chakraborty SS, Ward NP, Prieto-Farigua N, Falzone A, DeLany JP, Smith SR, Coen PM, DeNicola GM, Gardell SJ. Source of nicotinamide governs its metabolic fate in cultured cells, mice, and humans. Cell Rep. 2023 Mar 28;42(3):112218. doi: 10.1016/j.celrep.2023.112218. Epub 2023 Mar 9. PMID 36897780
- [Background] Kim LJ, Chalmers TJ, Madawala R, Smith GC, Li C, Das A, Poon EWK, Wang J, Tucker SP, Sinclair DA, Quek LE, Wu LE. Host-microbiome interactions in nicotinamide mononucleotide (NMN) deamidation. FEBS Lett. 2023 Sep;597(17):2196-2220. doi: 10.1002/1873-3468.14698. Epub 2023 Aug 9. PMID 37463842
- [Background] Xiao W, Wang RS, Handy DE, Loscalzo J. NAD(H) and NADP(H) Redox Couples and Cellular Energy Metabolism. Antioxid Redox Signal. 2018 Jan 20;28(3):251-272. doi: 10.1089/ars.2017.7216. Epub 2017 Jul 28. PMID 28648096
- [Background] Chellappa K, McReynolds MR, Lu W, Zeng X, Makarov M, Hayat F, Mukherjee S, Bhat YR, Lingala SR, Shima RT, Descamps HC, Cox T, Ji L, Jankowski C, Chu Q, Davidson SM, Thaiss CA, Migaud ME, Rabinowitz JD, Baur JA. NAD precursors cycle between host tissues and the gut microbiome. Cell Metab. 2022 Dec 6;34(12):1947-1959.e5. doi: 10.1016/j.cmet.2022.11.004. PMID 36476934
- [Background] Bhasin S, Seals D, Migaud M, Musi N, Baur JA. Nicotinamide Adenine Dinucleotide in Aging Biology: Potential Applications and Many Unknowns. Endocr Rev. 2023 Nov 9;44(6):1047-1073. doi: 10.1210/endrev/bnad019. PMID 37364580